CLINICAL TRIAL: NCT01924234
Title: Opioid Effects on Swallowing Comparing Younger and Elderly Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Johanna Savilampi, M.D., Region Örebro County
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JS004
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Pharyngeal Dysfunction; Pharyngeal Swallowing
Keywords: Remifentanil; Pharyngeal dysfunction; Subjective swallowing difficulties; Pulmonary aspiration
MeSH Terms: interventions — Morphine; Remifentanil; Powders; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- morphine (Active Comparator): Volunteers are given morphine injection
  Interventions: Drug: Morphine
- remifentanil (Active Comparator): Volunteers are given remifentanil infusion
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Morphine
  Other Names: ACT-code: N02AA01; Younger volunteers: injection 0.1 mg/kg; Elderly volunteers: injections 0.07 mg/kg
  Arms: morphine
Drug: Remifentanil
  Other Names: Ultiva; ATC-code: N01AH06; Powder for injection/ infusion fluid solution, 1 mg Infusion TCI 3 ng/ml 30 min ( 0,15 ug/kg/min)
  Arms: remifentanil

SUMMARY:
The purpose of the study is to determine whether remifentanil influence the pharyngeal phase of swallowing using using pressure and impedance recordings. The purpose is also to compare remifentanil to morphine and younger to elderly volunteers.

DETAILED DESCRIPTION:
Remifentanil and other opioids are widely used as anesthetic sedation during minor surgical procedures and as pain relief in postoperative patients when the patient is spontaneously breathing and the airway is not secured by endotracheal intubation. In a previous study (not yet published) we showed that remifentanil induce pulmonary aspiration in healthy volunteers and the aim of this study is to objectively determine weather remifentanil infusion in healthy volunteers influence the pharyngeal phase of swallowing. The purpose is also compare the effect of remifentanil to morphine and younger volunteers to elderly volunteers. To assess this question we are going to study 24 volunteers, 12 younger and 12 elderly, who are randomised to receive remifentanil infusion with target concentration 3 ng/ml during 30 minutes at one occasion and an injection of morphine (younger: 0.1 mg/kg, elderly 0.07 mg/kg) at the other. The volunteers are asked to swallow 10 ml normal saline several times both before and after opioid administration and pharyngeal motility is parallelly recorded using combined manometry and impedance catheter placed transnasally into to the pharyngo-esophageal segment. Any subjective swallowing difficulties are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 or 65 < year old healthy volunteers from both sexes.
* Have signed and dated Informed Consent.
* Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

* Pharyngoesophageal dysfunction
* Known history of cardiac, pulmonary or neurological disease
* Ongoing medication
* Allergies to or history of reaction to remifentanil, fentanyl analogues or other ingredients
* Pregnancy or breast feeding
* BMI > 30
* Previous participation in a medical clinical trial where opioid has been used or have during last 30 days participated in any other medicinal clinical trial or in a trial where follow-up in not complete.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pressure-Flow Variables measured by combined manometry and impedance system ( ManoScan 360) during pharyngeal swallowing | up to 30 minutes after opioidadministration (after start of remifentanil infusion or morphine injection)

SECONDARY OUTCOMES:
Subjective swallowing difficulties measured by 4-point scale | Variables are measured before (baseline) and 15 min and 30 minutes after opioidadministration (after start of remifentanil infusion or morphine injection)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Savilampi, M.D, Principal Investigator — Department of Anesthesiology and Intensive Care, Örebro University Hospital
Locations (1):
- Örebro University Hospital, Örebro, Sweden

REFERENCES:
- [Derived] Savilampi J, Omari T, Magnuson A, Ahlstrand R. Effects of remifentanil on pharyngeal swallowing: A double blind randomised cross-over study in healthy volunteers. Eur J Anaesthesiol. 2016 Sep;33(9):622-30. doi: 10.1097/EJA.0000000000000461. PMID 27191923